CLINICAL TRIAL: NCT01725243
Title: Carbetocin at Cesarean Delivery for Labor Arrest: A Dose Finding Study
Brief Title: Carbetocin at Cesarean Delivery for Labor Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-07
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin; failure to progress in labor
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Carbetocin 10mcg (Active Comparator): Carbetocin 10mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 20mcg (Active Comparator): Carbetocin 20mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 40mcg (Active Comparator): Carbetocin 40mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 60mcg (Active Comparator): Carbetocin 60mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 80mcg (Active Comparator): Carbetocin 80mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator): Carbetocin 100mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 120mcg (Active Comparator): Carbetocin 120mcg IV, once following delivery.
  Interventions: Drug: Carbetocin
- Carbetocin 140mcg (Active Comparator): Carbetocin 140mcg IV, once following delivery.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin IV, over 1 minute following delivery. Doses: 10, 20, 40, 60, 80, 100, 120 or 140mcg
  Other Names: Duratocin

SUMMARY:
In 2009, the Society of Obstetricians and Gynecologists Canada, which produces national clinical guidelines on important women's health issues, recommended that a bolus of carbetocin 100 mcg into your vein should be used at elective cesarean delivery instead of oxytocin infusion for the prevention of bleeding after you deliver your baby. Similar to oxytocin, carbetocin has side effects that are dose-related. Although 100 mcg has been the recommend dose, studies in nonlaboring women suggest that doses lower than 100 mcg may be used to achieve the same degree of uterine contractility with less side effects. So far, the ideal dose to be used in cesarean sections for labouring women who have failure to progress in labour (failure of your cervix to dilate adequately to 10cm or the baby's head not descending the birth canal) has not been determined. This study is designed to determine the minimum carbetocin dose required during cesarean delivery for 'failure to progress' to achieve the best effect.

DETAILED DESCRIPTION:
Post-partum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most common uterotonic drug used to prevent and treat PPH in North America, however, there are some limitations to its use. Oxytocin has a very short duration of action, which requires a continuous infusion to achieve sustained uterotonic activity. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recently recommended a single 100mcg dose of carbetocin at elective Cesarean delivery to promote uterine contraction and prevent post partum hemorrhage (PPH), in lieu of the more traditional oxytocin regimens. Carbetocin lasts 4 to 7 times longer than oxytocin, with a similar side effect profile and apparent greater efficacy rate.

The evidence reported for Carbetocin use in the literature has mostly been based upon low risk non-laboring patients undergoing elective cesarean deliveries. At present, only 2 studies have looked at the use of Carbetocin in low risk patients requiring emergency cesarean deliveries. The minimum effective dose (ED90) of carbetocin in laboring women has not been determined so far. Similar to oxytocin, the ED90 of Carbetocin is likely to be higher in laboring women undergoing Cesarean deliveries as compared to the non-laboring women, due to the effect of the desensitization phenomenon.

This study will be conducted as a prospective, randomized, up-down sequential allocation trial. The success or fail of a patient in the study will determine the dose given to future patients. Dosage will be increased for patients following a failed case, and kept the same for patients following successful cases. Following a successful case, there is also a 1 in 9 chance that the dose will be decreased for the next patient.

The results of this study will establish the minimum effective dose of carbetocin for uterine contraction at cesarean delivery for labor arrest. This will likely minimize unnecessary side effects caused by a large bolus dose of the drug, and improve quality and safety of patient care.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have given written informed consent to participate in this study.
* All patients planned for uncomplicated low transverse cesarean delivery secondary to labor arrest, under epidural anesthesia.
* ≥37 week pregnancy
* Singleton pregnancy
* Patients who have received oxytocin for at least 4 hours for labor augmentation
* ASA 1 or 2

Exclusion Criteria:

* Refusal or inability to obtain informed consent.
* All patients who claim allergy or hypersensitivity to oxytocin and carbetocin.
* Previous history of uterine atony or PPH
* Risk factors for PPH such as pre-eclampsia, polyhydramnios, uterine fibroids, bleeding diathesis and chorioamnionitis etc.
* Abnormal placental implantation (known or suspected)
* > 3 cesarean sections in the past
* Previous classic uterine incision
* Macrosomia - Estimated fetal weight > 4500g
* Hemoglobin < 100g/L
* Cesarean section under general anesthesia
* ASA 3 and 4 or patients with hepatic, renal, cardiac (eg. Coronary artery disease) and vascular disease
* Genital development problems (eg. Abnormal uterus, cervix, vagina, etc.)
* Uncontrolled hypotension or hypertension
* Uncontrolled diabetes
* Abnormal heart rhythms and bradycardia
* Drug abusers

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
need for additional uterotonics | 30 minutes
  need for additional uterotonics in the OR at the time of cesarean section based upon the assessment of unsatisfactory/indeterminate uterine tone in response to the single bolus of carbetocin.

SECONDARY OUTCOMES:
uterine tone | 10 minutes
  Incidence of satisfactory, unsatisfactory and indeterminate uterine tone at every minute for five minutes and at 10 minutes following the completion of the injection of carbetocin.
uterine tone | 2 hours
  Incidence of satisfactory, unsatisfactory/ indeterminate uterine tone as determined by the obstetrician/nurse after trans-abdominal palpation of the uterus in PACU within 2 hours of delivery of the placenta
need for additional uterotonic | 24 hours
  Need for delayed additional uterotonics within 24 hours after delivery outside the OR.
Blood loss | 24 hours
  Estimated blood loss will be calculated using blood results prior to the cesarean delivery and 24 hours post-delivery.
side effects | 2 hours
  Any of the following will be noted up to 2 hours post delivery: systolic blood pressure < 80% of pre-delivery values, tachycardia > 30% pre-delivery levels, bradycardia < 30% pre-delivery levels, other dysrhythmias, nausea, vomiting, chest pain, shortness of breath, headache, flushing, others

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nguyen-Lu N, Carvalho JC, Farine D, Seaward G, Ye XY, Balki M. Carbetocin at Cesarean delivery for labour arrest: a sequential allocation trial to determine the effective dose. Can J Anaesth. 2015 Aug;62(8):866-74. doi: 10.1007/s12630-015-0375-2. Epub 2015 Apr 10. PMID 25860126